CLINICAL TRIAL: NCT01691846
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Phase III Study to Assess the Efficacy, Safety and Tolerability of Aleglitazar Plus Metformin Combination Therapy Compared With Placebo Plus Metformin in Patients With T2D Inadequately Controlled With Metformin Monotherapy
Brief Title: A Study of Aleglitazar in Combination With Metformin in Patients With Type 2 Diabetes Mellitus Who Are Inadequately Controlled With Metformin Alone
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BC28035
Record Dates: First submitted 2012-09-20; First posted 2012-09-25 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- aleglitazar (Experimental)
  Interventions: Drug: aleglitazar+metformin
- placebo (Placebo Comparator)
  Interventions: Drug: placebo+metformin

INTERVENTIONS:
Drug: aleglitazar+metformin — 150 mcg aleglitazar given orally once a day for 26 weeks. Patients will continue on their existing dose and regimen of metformin (≥ 1500 mg/day or individual maximally tolerated dose)
  Arms: aleglitazar
Drug: placebo+metformin — Oral doses of matching placebo once a day for 26 weeks. Patients will continue on their existing dose and regimen of metformin (≥ 1500 mg/day or individual maximally tolerated dose)
  Arms: placebo

SUMMARY:
This multicenter, randomized, double-blind, placebo-controlled study will assess the efficacy, safety and tolerability of aleglitazar plus metformin combination therapy compared with placebo plus metformin in patients with type 2 diabetes mellitus who are inadequately controlled with metformin monotherapy. Patients will be randomized to receive oral doses of 150 mcg aleglitazar once daily or placebo. The anticipated time on study treatment is 26 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/=18 years of age
* Diagnosis of diabetes mellitus type 2
* Patients treated with stable metformin monotherapy for at least 12 weeks prior to screening
* HbA1c >/=7% and </=9.5% at screening or within 4 weeks prior to screening and at pre-randomization visit
* Fasting plasma glucose </=240 mg/dL at pre-randomization visit
* Agreement to maintain diet and exercise habits during the study

Exclusion Criteria:

* Patients with Type 1 diabetes mellitus, secondary diabetes, diabetes resulting from pancreatic injury, or acute metabolic diabetic complications within the past 6 months
* Any previous treatment with thiazolidinedione or a dual PPAR agonist
* Any body weight lowering or lipoprotein-modifying therapy within 12 weeks prior to screening (except stable dose of statin)
* Symptomatic congestive heart failure classified as New York Heart Association class II-IV at screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2012-10; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in hemoglobin HbA1c | From baseline to week 26

SECONDARY OUTCOMES:
Change in lipid profile | From baseline to week 26
Change from baseline in fasting plasma glucose | From baseline to week 26
Responder rate as defined of hemoglobin HbAc1 <7.0% (<6.5%) | From baseline to week 26
Change from baseline in homeostatic index of insulin sensitivity (HOMA-IS) | From baseline to week 26
Change from baseline in homeostatic index of beta cell function (HOMA-BCF) | From baseline to week 26
Safety: incidence of adverse events | 30 weeks (26 weeks treatment and 4 weeks follow-up)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (31):
- United States (22):
  - Chino, California
  - Hawaiian Gardens, California
  - Los Angeles, California
  - Santa Ana, California
  - Thousand Oaks, California
  - West Hills, California
  - Kissimmee, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Avon, Indiana
  - Bethesda, Maryland
  - Springfield, Missouri
  - Toms River, New Jersey
  - Altoona, Pennsylvania
  - Beaver, Pennsylvania
  - Morrisville, Pennsylvania
  - Scranton, Pennsylvania
  - Tipton, Pennsylvania
  - Knoxville, Tennessee
  - Dallas, Texas
  - Richmond, Virginia
  - Spokane, Washington
- Argentina (3):
  - Buenos Aires
  - Caba
  - Rosario
- Mexico (6):
  - Cuernavaca
  - Culiacán
  - Guadalajara
  - Mexico City
  - Pachuca
  - Tampico